CLINICAL TRIAL: NCT02637193
Title: A Single Center, Three Period, Randomized, Three-way Crossover, Double-blind Placebo And Moxifloxacincontrolled Study To Assess The Effects Of Effexor Xr On Cardiac Repolarization In Healthy Adult Subjects
Brief Title: A Study to Assess The Effects Of Effexor XR On Cardiac Repolarization In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: B2411360; TQTC (Other: Alias Study Number)
Record Dates: First submitted 2015-11-24; First posted 2015-12-22 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2018-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Venlafaxine Hydrochloride; Bulk Drugs; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Venlafaxine (Experimental): Maximum dose of 450 mg/day (225 mg BID given at approximately 12 hours apart) Venlafaxine, dose titrated from a starting single dose (QD) of 75 mg venlafaxine in the morning of Days 1 and 2, followed by BID escalating doses administered on Days 3 through 10, followed by 450 mg/day (BID) on Days 11 through 13, and on Day 14 only the morning dose of 225 mg will be administered, then 3 days (Days 15, 16 and 17) of down titration
  Interventions: Drug: Venlafaxine
- Moxifloxacin (Active Comparator): 400 mg single dose of moxifloxacin (Avelox®) administered on Day 14
  Interventions: Drug: Moxifloxacin
- Drug -- placebo (Placebo Comparator): Placebo administered on Days 1 through 13 and on Days 15 to 17
  Interventions: Drug: Drug - placebo

INTERVENTIONS:
Drug: Venlafaxine — Multiple doses of Venlafaxine for 14 days plus 3 days of down titration
  Other Names: Active drug
  Arms: Venlafaxine
Drug: Moxifloxacin — 400 mg single dose moxifloxacin
  Other Names: Positive control
  Arms: Moxifloxacin
Drug: Drug - placebo — Placebo administered for 16 days
  Other Names: Placebo control
  Arms: Drug -- placebo

SUMMARY:
The purpose of this study is to demonstrate a lack of effect of venlafaxine (Effexor XR) on QTc intervals relative to time matched placebo in healthy volunteers

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blinded, placebo- and moxifloxacin-controlled, 3 period, 6-sequence, 3 treatment (venlafaxine and placebo blinded; moxifloxacin open label), 3-way crossover thorough QT (TQT) study of the effects of venlafaxine on cardiac repolarization in approximately 54 healthy subjects

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy female subjects and/or male subjects who at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Based on CYP2D6 genotyping, the subject is required to be classified as a CYP2D6 extensive metabolizer (EM).

Main Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug screen.
4. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study medication (whichever is longer).
6. Screening supine blood pressure > 140 mm Hg (systolic) or > 90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >140 mm Hg (systolic) or >90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
7. Screening supine 12 lead ECG demonstrating QTcF >450 msec or a QRS interval >120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.
8. Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children and female subjects of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product or longer based upon the compound's half-life characteristics.
9. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication.
10. As an exception, acetaminophen/paracetamol may be used at doses of less than 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.

    Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of study medication.
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
12. History of sensitivity to heparin or heparin induced thrombocytopenia.
13. History of known QTc prolongation or ECG abnormalities.
14. Individuals with known hypersensitivity reactions to venlafaxine, desvenlafaxine or SSRI (Selective serotonin reuptake inhibitors) or SNRI (Selective serotonin and norepinephrine reuptake inhibitors).
15. Individuals with a known hypersensitivity to moxifloxacin or quinolones.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Postdose QTcF (Fridericia's correction) intervals | 0 to 24 hours

SECONDARY OUTCOMES:
Averse events, vital signs, physical examinations and abnormal laboratory for safety assessments (safety and tolerability) | Through the study completion, an average of 3 months
Relationship between QTc prolongation and the measured venlafaxine/desvenlafaxine plasma concentration | 0 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2411360&StudyName=A%20Single%20Center%2C%20Three%20Period%2C%20Randomized%2C%20Three-way%20Crossover%2C%20Double-blind%20Placebo%20And%20Moxifloxacincontrolled%20Study%20To%20Assess%20The%20Effects%20Of%20Effexor%20Xr%20On%20Cardiac%20Repolarization%20In%20Healthy%20Adult%20Subjects